CLINICAL TRIAL: NCT05978050
Title: Nimotuzumab Combined With Paclitaxel as Second-line Treatment for Recurrent Metastatic Gastric or Esophagogastric Junction Adenocarcinoma With EGFR Over-expression: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial
Brief Title: Nimotuzumab Combined With Paclitaxel for Recurrent Metastatic Gastric or Esophagogastric Junction Adenocarcinoma
Acronym: NOTABLE-307
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPL-Nim-GC-3001
Record Dates: First submitted 2023-07-20; First posted 2023-08-07 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Gastric or Esophagogastric Junction Adenocarcinoma
MeSH Terms: interventions — nimotuzumab; Paclitaxel; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nimotuzumab (Experimental): Participants received nimotuzumab injection 600 mg for the first time, followed by 400 mg once a week until disease progression or inability to tolerate or withdrawal from the trial; At the same time, in combination with paclitaxel 80 mg/m2, it was administered on days 1, 8 and 15 of each treatment cycle (4 weeks) until the disease progressed or could not be tolerated or withdrew from the trial.
  Interventions: Drug: nimotuzumab plus paclitaxel
- placebo (Placebo Comparator): Participants received placebo 600 mg for the first time, followed by 400 mg once a week until disease progression or inability to tolerate or withdrawal from the trial; At the same time, in combination with paclitaxel 80 mg/m2, it was administered on days 1, 8 and 15 of each treatment cycle (4 weeks) until the disease progressed or could not be tolerated or withdrew from the trial.
  Interventions: Drug: placebo plus paclitaxel

INTERVENTIONS:
Drug: nimotuzumab plus paclitaxel — Nimotuzumab injection: 50mg/10ml/stick Paclitaxel: 30mg/5ml/stick
  Other Names: Combined with chemotherapy
  Arms: nimotuzumab
Drug: placebo plus paclitaxel — placebo: 50mg/10ml/stick Paclitaxel: 30mg/5ml/stick
  Other Names: chemotherapy alone
  Arms: placebo

SUMMARY:
In order to evaluate the efficacy and safety of nimotuzumab combined with paclitaxel as second-line treatment for recurrent metastatic gastric or esophagogastric junction adenocarcinoma with EGFR over-expression, investigators performed a randomized, double-blind, placebo-controlled phase III clinical trial. Patients will be randomized (1:1) to receive nimotuzumab plus paclitaxel in the experimental group and placebo plus paclitaxel in the control group. The primary endpoint of this study was OS, and according to the results of the RAINBOW-Asia gastric cancer phase III clinical study, the mOS of paclitaxel single-agent second-line treatment for gastric cancer was 7.92 months, assuming that the mOS increased to 10.92 months after the addition of nimotuzumab, Using the survival module in the PASS15 software, the two-sided test level was set α=0.05, β=0.20, enrolled for 2 years, followed up for 1.5 years, the dropout rate was 5%, the sample size including interim analysis was 354 cases. The secondary endpoints are progression-free survival (PFS), objective response rate (ORR), duration of response (DOR), disease control rate (DCR), patient reported outcome (PRO), and safety.

DETAILED DESCRIPTION:
Study design:

This study is a prospective, randomized, double-blind, placebo-controlled trial designed to evaluate the efficacy and safety of nimotuzumab combined with paclitaxel as second-line treatment for recurrent metastatic gastric or esophagogastric junction adenocarcinoma with EGFR over-expression.A total of 354 patients with recurrent metastatic gastric or esophagogastric junction adenocarcinoma with EGFR over-expression are expected to be enrolled. Patients will be randomized (1:1) to receive nimotuzumab (600 mg for the first dose, then 400 mg, weekly) plus paclitaxel (80 mg/m2, on day 1, 8 and 15, every 4 weeks as a cycle) in the experimental group and placebo plus paclitaxel (same as experimental group) in the control group. The study will be randomized by stratified block randomization, stratification factors included ECOG PS (0 vs. 1), first-line immunotherapy (yes vs. no), and EGFR expression status (IHC 2+ vs. 3+). Treatment will continue until disease progression, intolerance, or patient withdrawal from the trial, and each patient will be followed up until death, loss to follow-up, or the end of study.

Quality Assurance plan： According to the GCP's guidelines, sponsors are responsible for using and maintaining quality assurance and quality control systems in accordance with the corresponding standard operating procedures (SOPs). The sponsor or sponsor's representative shall conduct quality control at every stage of data processing to ensure the accuracy, consistency, completeness and reliability of the data. In addition, the sponsor or its representative, the appropriate regulatory body, may conduct audits and/or inspections of the research process. During audits and/or regulatory inspections, authorized sponsor representatives and relevant regulatory authorities have access to all research-related documents.

Data checks:

Investigators should collect complete participant data as required by the protocol, recorded in the original record. This study will use an electronic data acquisition (EDC) system, and the library builder will build an electronic database according to the plan, set up the corresponding logic verification, and data management personnel will conduct data verification according to the corresponding verification plan.

Source data verification:

The research data will be entered into the eCRF by the researcher or authorized research center staff. Investigators review the data to ensure the accuracy of all data entered into the eCRF. The eCRF will be reviewed by the Inspector and assessed for completeness and consistency, and the Auditor will compare the eCRF with the original documentation to ensure consistency of critical data. All data entry, correction and modification will be the responsibility of the researcher or its designee, and the supervisor will not have this authority. The data in the eCRF is submitted to the data server, and any changes to the data will be recorded in the audit track, that is, the reason for the change, the operator account number, the modification time and date will be recorded. If there is a data challenge, the monitor, medical or data management personnel will issue the challenge in the EDC according to the corresponding verification plan, and the research center staff will be responsible for answering the question, and conduct data verification from multiple parties and angles to ensure data quality. After all data has been entered into the EDC in its entirety, the monitor has completed the SDV on all data in the EDC, the medical and data administrator has completed the review of all data in the EDC, and all challenges have been closed, the data administrator freezes the data.

Data dictionary:

The combined medication and medical history will be encoded using the Anatomical, Therapeutic, and Chemical Taxonomy of Drugs (ATC 2021 and above) and the Regulatory Activities Medical Dictionary (MedDRA V24.0 and above), respectively.

Standard Operating Procedures:

Informed consent approved by the Independent Ethics Committee (IEC)/Institutional Review Board (IRB) must be obtained prior to carrying out any research-specific procedures. Potentially eligible subjects will be screened within 4 weeks prior to the first dose, and after qualified subject screening, they will be enrolled through an interactive web response system (IWRS). Investigators should collect complete participant data (e.g., laboratory tests, vital signs, physical examination, electrocardiogram, imaging tests, adverse effects, quality of life assessment scale evaluation, etc.) as required by the protocol and record them in the original record.

Investigators are required to submit a completed eCRF for each participant enrolled in the study. Study numbers and subject numbers submitted with the eCRF should be carefully verified and all private information (including subject names) removed or rendered illegible to protect subject privacy. When researching data entry into eCRF, the system will automatically add the identity of the data entry user by the ID of the login user. The investigator proves that it has reviewed the record through an electronic signature record and guarantees the accuracy of the data in the record. After all data in the EDC is reviewed and all doubts have been closed, the data is locked and analyzed.

Adverse events were monitored throughout the study and it was the responsibility of the investigator to document all AEs observed during the study. From the beginning of the subject's signing of informed consent to 30 days after the last dose of the investigational drug, all AEs, regardless of severity and causal relationship with the investigational drug, need to be recorded in the original data and the corresponding AE page in the eCRF. According to the relevant regulations of ICH and China GCP (2020 edition), during this study, investigators should complete the SAE report form provided by the sponsor and report to the sponsor in writing within 24 hours after learning of SAE or relevant new follow-up information.

Sample size:

The primary endpoint of this study was OS, and according to the results of the RAINBOW-Asia gastric cancer phase III clinical study, the mOS of paclitaxel single-agent second-line treatment for gastric cancer was 7.92 months, assuming that the mOS increased to 10.92 months after the addition of nimotuzumab, and an interim analysis was set up during the trial. Using the survival module in the PASS15 software, the two-sided test level was set α=0.05, β=0.20, enrolled for 2 years, followed up for 1.5 years, the dropout rate was 5%, the single-stage sample size was 354 cases, and the required sample size for each group was 177.

Plan for missing data:

For participants who had not reported death at the time of analysis, the last known surviving follow-up date was used as the censoring date. For subjects who have not yet progressed, the date of the last radiographic evaluation is used as the date of censoring. For participants who had not undergone tumour assessment after baseline, the date of randomisation was used as the date of censoring.

Statistical analysis plan:

The main overall survival (OS) analysis will be performed when 306 death events occur, optimality test and blind sample size adjustment will be performed when 50% of death events occur.

The primary endpoint of this study was mOS. OS is the time between the date of randomization and death from any cause. A stratified log-rank test was used to compare OS in the nilotuzumab plus paclitaxel and placebo plus paclitaxel group at a bilateral significance level of 0.05. The Kaplan-Meier (KM) method was used to estimate the OS of each treatment group, and the Kaplan-Meier curve was plotted to show the survival difference description. Efficacy estimates of OS will be expressed by risk ratios (HR) estimated by the hierarchical Cox proportional hazards model and their 95% confidence intervals.

Secondary endpoints: PFS, ORR, DOR, DCR，PRO and safety. The Kaplan-Meier (KM) method was used to estimate the PFS of each treatment group, and the Kaplan-Meier curve was plotted to show the difference description. The stratification factors are the same as for OS analysis. Efficacy estimates of PFS will be expressed by risk ratios (HR) estimated by the hierarchical Cox proportional hazards model and their 95% confidence intervals. The Clopper-Pearson exact probability method was used to calculate the ORR and DCR estimates and their 95% confidence intervals for each treatment group, respectively. The Cochran-Mantel-Haenszel (CMH) method was used to calculate the odds ratio and its 95% confidence interval and p. The stratification factors used in the CMH test are the same as in the OS analysis. If the number of objective remission or disease control cases is insufficient to support the CMH test, stratified precision testing is considered and precise confidence intervals for odds ratios are calculated. DOR is only available for participants with objective response (CR/PR) for descriptive analysis of TOR. Results will be shown using the Kaplan-Meier method for each treatment group to estimate the median DOR and the distribution curve.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-75 years old (including boundary value), male or female;
* 2. The physical status score ECOG is 0-1;
* 3. Histopathologically or cytologically confirmed gastric or esophagogastric junction adenocarcinoma;
* 4. Recurrent metastatic disease, previous treatment with first-line standard chemotherapy regimens (including platinum-containing and/or fluorouracil regimens) (recurrence or metastasis during adjuvant therapy or within 6 months after completion is considered first-line therapy), or received anti-HER2 therapy, or received immunotherapy, and has been confirmed by the investigator or has a clear disease progression in the medical history;
* 5. At least one evaluable tumor lesion according to the RECIST version 1.1 evaluation criteria;
* 6. Detection of primary or metastatic lesions during the screening period (when multiple specimens exist at the same time, the bulk specimen is preferred over the biopsy specimen, and the metastasis is preferred over the primary lesion) tissue is determined to be EGFR high expression (IHC2+ or IHC3+);
* 7. Estimated survival≥ 12 weeks;
* 8. Have proper organ function, defined as:Total bilirubin ≤ 1.5 times the upper normal limit (ULN); glutamyltransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5 times ULN in the absence of liver metastases; ALT or AST ≤ 5 times ULN in the presence of liver metastases;Serum creatinine level≤ 1.5 times ULN; neutrophil count ≥1.5×109/L; WBC count≥ 3.0×109/L; platelets≥ 100×109/L; Hemoglobin≥ 90g/L;
* 9. Patients of childbearing age and their spouses are willing to use contraception;
* 10. Women of potential fertility have negative serum hCG within 72 hours prior to randomization (postmenopausal women with amenorrhea for at least 12 months are considered infertile, and women who are known to have undergone tubal ligation are not required to undergo a pregnancy test);
* 11. The subject understands and complies with the study process, voluntarily participates, and signs the informed consent form.

Exclusion Criteria:

* 1. Received the following treatments before this study:

  1. The disease has progressed after previous paclitaxel chemotherapy or molecular targeted drug (anti-EGFR antibody) treatment, or received paclitaxel chemotherapy or molecular targeted drug (anti-EGFR antibody) treatment within 4 weeks before randomization;
  2. Within 4 weeks before randomization or participating in other therapeutic/intervention clinical trials or receiving combined treatment prohibited by the protocol;
* 2. Received major surgical treatment, incision biopsy (such as laparotomy) or obvious traumatic injury within 4 weeks before randomization;
* 3. Brain metastases or meningeal metastases;
* 4. Has a history of malignant tumors other than gastric adenocarcinoma or esophagogastric junction adenocarcinoma (except for cured cervical carcinoma in situ or skin basal cell carcinoma and other malignant tumors that have been cured for 5 years);
* 5. Known to have suffered from severe bleeding disorders (such as severe gastrointestinal bleeding) and vasculitis within 3 months before randomization;
* 6. Known to be accompanied by other serious diseases, including but not limited to:

  1. Refractory congestive heart failure (NYHA classification III or IV, see Appendix 2), unstable angina, poorly controlled arrhythmia, uncontrolled moderate or high blood pressure (SBP>160mmHg or DBP>100mmHg );
  2. Uncontrolled diabetes;
  3. Mental illness that affects informed consent and/or protocol compliance;
  4. There are serious diseases that other researchers believe are not suitable for participating in this study;
* 7. Known allergies or contraindications to anti-EGFR antibody preparations, paclitaxel and other components;
* 8. Patients who have previously used immune checkpoint inhibitors (such as anti-PD-1, anti-PD-L1, anti-CTLA-4 antibodies), such as the following adverse events related to immune checkpoint inhibitors and have not recovered to grade 1 And below, not suitable for inclusion: Grade ≥3 ocular adverse events, abnormal liver function in line with Hy's Law standard adverse events, ≥3 neurological toxicity, ≥3 grade colitis, ≥3 grade renal toxicity;
* 9. Those who are known to have third space effusion (including a large amount of pleural effusion or ascites) that cannot be controlled by drainage or other methods;
* 10. Known NCI CTC grade 2-4 peripheral neuropathy;
* 11. Known history of primary or secondary immunodeficiency or current active primary or secondary immunodeficiency;
* 12. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA ≥ 1000 IU/ml or hepatitis C virus (HCV) RNA positive (inactive hepatitis B surface antigen carriers, treated And stable hepatitis B patients [HBV DNA <1000 IU/ml and cured hepatitis C patients can be selected]); Treponema pallidum antibody positive or human immunodeficiency virus antibody positive or any uncontrolled infection By;
* 13. Women of childbearing age who are pregnant, breast-feeding, planning to become pregnant, or who have not taken reliable birth control measures and men in the sexually active period who are unwilling to take birth control measures during the study period and within 3 months after the last medication, and during the above-mentioned specified time Sperm donors;
* 14. Any medical, psychiatric or other condition or situation that the investigator believes that the subject's participation in this clinical research may have a negative impact on the safety of the subject or the reliability of the research data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 354 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | through study completion, an average of 18 months
  The time between the date of randomization and death from any cause .

SECONDARY OUTCOMES:
progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  The time between the date of randomization and the date of PD or death when PD was first recorded, whichever occurs first
objective response rate | Assessment is performed every 4 weeks for the first 3 months, every 8 weeks to 12 months thereafter, and every 3 months thereafter until disease progression ,assessed up to 12 months
  The optimal total response (BOR) is the incidence of complete response (CR) or partial response (PR).
DCR | Assessment is performed every 4 weeks for the first 3 months, every 8 weeks to 12 months thereafter, and every 3 months thereafter until disease progression,assessed up to 12 months
  CR+PR+SD

CONTACTS AND LOCATIONS:
Overall Officials: ruihua Xu, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- National Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No